CLINICAL TRIAL: NCT03794518
Title: Effect of Combination Therapy With Dapagliflozin Plus Low Dose Pioglitazone on Hospitalization Rate in Patients With Heart Failure and Preserved Left Ventricular Ejection Fraction
Brief Title: Effect of Dapagliflozin Plus Low Dose Pioglitazone on Hospitalization Rate in Patients With HF and HFpEF
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRGC-04-SI-17-116
Record Dates: First submitted 2018-08-01; First posted 2019-01-07 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2018-07

CONDITIONS: Risk Reduction
MeSH Terms: conditions — Risk Reduction Behavior | interventions — Pioglitazone

STUDY DESIGN:
Intervention Model Description: Pioglitazone (15 mg) and dapagliflozin (10mg) vs Placebo
Who Masked: Participant
Masking Description: Random process
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pioglitazone Plus dapaglifliozin (Experimental): Pioglitazone 15mg and dapaglifliozin 10mg together in T2DM patients having HF and HFpEF conditions
  Interventions: Drug: Pioglitazone Plus dapaglifliozin
- Placebo (Placebo Comparator): Beta blockers, ACEI, ARB, and aldosterone
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone Plus dapaglifliozin — Pioglitazone Plus dapaglifliozin
  Arms: Pioglitazone Plus dapaglifliozin
Drug: Placebo — (Beta blockers, ACEI, ARB, and aldosterone )
  Arms: Placebo

SUMMARY:
The prevalence of type 2 diabetes mellitus (T2DM) in Qatar and nations worldwide has increased in recent decades into epidemic proportions. Cardiovascular (CVD) disease is the leading cause of death in T2DM patients. Approximately 80% of T2DM patients will die because of CV cause. Congestive heart failure (CHF) is a major cause of CV death in T2DM, and it also is responsible for significant morbidity and health care expenditure due to high rate of hospitalization for heart failure.

DETAILED DESCRIPTION:
Community based studies have demonstrated similar prevalence of HF with reduced ejection fraction (HFpEF) and HF with reduced LV function (HFrEF) in patients hospitalized for CHF. Moreover, the prevalence of HFrEF is declining over the past two decades, whereas that of HFpEF is progressively increasing. Progressive increase in obesity and T2DM prevalence is likely among the principal factors responsible for the steady increase in HFpEF prevalence.

The aims of the present study are to examine whether therapies that correct the myocardial metabolic abnormalities present in subjects with T2DM and diastolic dysfunction improve myocardial diastolic dysfunction and reduce the rate of hospitalizations in patients with HFpEF

The primary objective of the study is to examine the effect of combination therapy with pioglitazone (15 mg) plus dapagliflozin (10 mg) versus placebo on hospitalization for heart failure in patients with HFpEF.

Eligible subjects, who consent for participating in the study, will be seen by the study coordinator. Medical history and physical examination will be performed. Each subject will receive the following measurements:

Medical history and physical examination including weight, height, waist, blood pressure and pulse.

Blood tests:

Screening: CBC, Blood chemistry, fasting plasma glucose concentration, HbA1c, renal and liver function, lipid profile, TSH, serum iron, iron biding capacity and ferritin.

Plasma metabolites: ketone, lactate, bicarbonate, venous PH and plasma free fatty acid.

Hormones: insulin, C-peptide, glucagon, NT proBNP, angiotensin II, plasma renin activity, and aldosterone.

Inflammatory markers: adiponectin, hsCRP, IL-2, IL-6 and IL-12, F2-isoprostane, oxidized LDL.

Vascular Measurements: Measurement of pulse wave velocity, and central aortic pulse pressure, with sphygmocor.

Measurement of total body fat mass with Bioimpedence. Echocardiography

Patients will be consented on the day of discharge or during the outpatient visit in the Cardiology Clinic. Consented patients will be referred to the CRC within one week to perform the echocardiography and vascular measurements. Patients will be asked to come to CRC after overnight fast and blood samples will be drawn for the above mentioned blood tests, after which echocardiography and vascular measurements will be performed.

Randomization and Intervention:

After completing the baseline studies, patients will be randomized into two groups to receive in a double blind fashion:

Group 1: combination of pioglitazone plus dapagliflozin, or Group 2: Placebo (Beta blockers, ACEI, ARB, and aldosterone )

Patients in both groups will be matched for age, gender, BMI, HbA1c, systolic BP and LVEF. Randomization will be made by the pharmacist at the Heart Hospital and the randomization code will be maintained at the hospital pharmacy. Patients will be randomized in blocks of 4 while the group means are matched for the above parameters

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of type 2 diabetes according to the ADA criteria.
2. Drug naïve or on stable dose of antidiabetic therapy (oral agents and/or insulin) for 3 months preceding recruitment.
3. Hospitalized for HFpEF (defined as hospitalization require intravenous diuresis) in the 6 months preceding recruitment.
4. eGFR >60 ml/min
5. LVEF >50%
6. Presence of LV diastolic dysfunction in echocardiography

We have limited the inclusion criteria in the present study to T2DM patients with HFpEF and evidence of diastolic dysfunction by echocardiography in order to select a homogenous group of HFpEF patients with similar etiology, likely "metabolic HFpEF". We believe that this subgroup of HFpEF will benefit most from treatment with low dose pioglitazone (15 mg) plus dapagliflozin (10 mg).

Exclusion Criteria:

1. Treatment with pioglitazone or SGLT2 inhibitor in the 3 months prior to recruitment.
2. eGFR < 60 ml/min
3. LVEF <50%;
4. Valvular heart disease, ASD, VSD
5. Chronic lung disease
6. Cancer
7. diabetes mellitus type 1
8. patients with acute coronary syndrome, stroke or transient ischemic attack in the preceding 6 months
9. pregnancy or lactation period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 648 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Time to first hospitalization for heart failure after starting intervention | 3 years
  Hospitalization for heart failure will be defined as a hospitalization >24 hours requiring intravenous diuretic infusion.

SECONDARY OUTCOMES:
Number of all cause mortality | 3 years
  Composite outcome comprised of total mortality, incidence of acute coronary syndrome and non fatal CVA

CONTACTS AND LOCATIONS:
Overall Officials: Nidal Asaad, MD, Principal Investigator — Heart Hospital, HMC, Doha, Qatar
Locations (1):
- Heart Hospital, Hamad Medical Coorporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alharbi NS, Almutari R, Jones S, Al-Daghri N, Khunti K, de Lusignan S. Trends in the prevalence of type 2 diabetes mellitus and obesity in the Arabian Gulf States: systematic review and meta-analysis. Diabetes Res Clin Pract. 2014 Nov;106(2):e30-3. doi: 10.1016/j.diabres.2014.08.019. Epub 2014 Sep 6. PMID 25241351
- [Result] Shaw JE, Sicree RA, Zimmet PZ. Global estimates of the prevalence of diabetes for 2010 and 2030. Diabetes Res Clin Pract. 2010 Jan;87(1):4-14. doi: 10.1016/j.diabres.2009.10.007. Epub 2009 Nov 6. PMID 19896746
- [Result] American Diabetes Association. 9. Cardiovascular Disease and Risk Management. Diabetes Care. 2017 Jan;40(Suppl 1):S75-S87. doi: 10.2337/dc17-S012. No abstract available. PMID 27979896
- [Result] Bahrami H, Bluemke DA, Kronmal R, Bertoni AG, Lloyd-Jones DM, Shahar E, Szklo M, Lima JA. Novel metabolic risk factors for incident heart failure and their relationship with obesity: the MESA (Multi-Ethnic Study of Atherosclerosis) study. J Am Coll Cardiol. 2008 May 6;51(18):1775-83. doi: 10.1016/j.jacc.2007.12.048. PMID 18452784
- [Result] Kannel WB, Hjortland M, Castelli WP. Role of diabetes in congestive heart failure: the Framingham study. Am J Cardiol. 1974 Jul;34(1):29-34. doi: 10.1016/0002-9149(74)90089-7. No abstract available. PMID 4835750
- [Result] Nichols GA, Gullion CM, Koro CE, Ephross SA, Brown JB. The incidence of congestive heart failure in type 2 diabetes: an update. Diabetes Care. 2004 Aug;27(8):1879-84. doi: 10.2337/diacare.27.8.1879. PMID 15277411
- [Result] Gustafsson I, Brendorp B, Seibaek M, Burchardt H, Hildebrandt P, Kober L, Torp-Pedersen C; Danish Investigatord of Arrhythmia and Mortality on Dofetilde Study Group. Influence of diabetes and diabetes-gender interaction on the risk of death in patients hospitalized with congestive heart failure. J Am Coll Cardiol. 2004 Mar 3;43(5):771-7. doi: 10.1016/j.jacc.2003.11.024. PMID 14998615
- [Result] Pfeffer MA, Braunwald E, Moye LA, Basta L, Brown EJ Jr, Cuddy TE, Davis BR, Geltman EM, Goldman S, Flaker GC, et al. Effect of captopril on mortality and morbidity in patients with left ventricular dysfunction after myocardial infarction. Results of the survival and ventricular enlargement trial. The SAVE Investigators. N Engl J Med. 1992 Sep 3;327(10):669-77. doi: 10.1056/NEJM199209033271001. PMID 1386652
- [Result] Owan TE, Hodge DO, Herges RM, Jacobsen SJ, Roger VL, Redfield MM. Trends in prevalence and outcome of heart failure with preserved ejection fraction. N Engl J Med. 2006 Jul 20;355(3):251-9. doi: 10.1056/NEJMoa052256. PMID 16855265
- [Result] Shah SJ, Katz DH, Selvaraj S, Burke MA, Yancy CW, Gheorghiade M, Bonow RO, Huang CC, Deo RC. Phenomapping for novel classification of heart failure with preserved ejection fraction. Circulation. 2015 Jan 20;131(3):269-79. doi: 10.1161/CIRCULATIONAHA.114.010637. Epub 2014 Nov 14. PMID 25398313
- [Result] Johnsson K, Johnsson E, Mansfield TA, Yavin Y, Ptaszynska A, Parikh SJ. Osmotic diuresis with SGLT2 inhibition: analysis of events related to volume reduction in dapagliflozin clinical trials. Postgrad Med. 2016 May;128(4):346-55. doi: 10.1080/00325481.2016.1153941. Epub 2016 Mar 2. PMID 26878357
- [Result] Liu C, Liu T, Li G. Pioglitazone may offer therapeutic advantages in diabetes-related atrial fibrillation. Int J Cardiol. 2013 Sep 30;168(2):1603-5. doi: 10.1016/j.ijcard.2013.01.037. Epub 2013 Feb 12. No abstract available. PMID 23414743
- [Result] Liu B, Wang J, Wang G. Beneficial effects of pioglitazone on retardation of persistent atrial fibrillation progression in diabetes mellitus patients. Int Heart J. 2014;55(6):499-505. doi: 10.1536/ihj.14-107. Epub 2014 Oct 14. PMID 25310928
- [Result] Sulaiman K, Panduranga P, Al-Zakwani I, Alsheikh-Ali AA, AlHabib KF, Al-Suwaidi J, Al-Mahmeed W, AlFaleh H, Elasfar A, Al-Motarreb A, Ridha M, Bulbanat B, Al-Jarallah M, Bazargani N, Asaad N, Amin H. Clinical characteristics, management, and outcomes of acute heart failure patients: observations from the Gulf acute heart failure registry (Gulf CARE). Eur J Heart Fail. 2015 Apr;17(4):374-84. doi: 10.1002/ejhf.245. Epub 2015 Mar 4. PMID 25739882
- [Result] Abdul-Ghani M, Migahid O, Megahed A, Adams J, Triplitt C, DeFronzo RA, Zirie M, Jayyousi A. Erratum. Combination Therapy With Exenatide Plus Pioglitazone Versus Basal/Bolus Insulin in Patients With Poorly Controlled Type 2 Diabetes on Sulfonylurea Plus Metformin: The Qatar Study. Diabetes Care 2017;40:325-331. Diabetes Care. 2017 Aug;40(8):1134. doi: 10.2337/dc17-er08d. Epub 2017 Jun 14. No abstract available. PMID 28615237
- [Result] Abdul-Ghani M, Migahid O, Megahed A, Adams J, Triplitt C, DeFronzo RA, Zirie M, Jayyousi A. Combination Therapy With Exenatide Plus Pioglitazone Versus Basal/Bolus Insulin in Patients With Poorly Controlled Type 2 Diabetes on Sulfonylurea Plus Metformin: The Qatar Study. Diabetes Care. 2017 Mar;40(3):325-331. doi: 10.2337/dc16-1738. Epub 2017 Jan 17. PMID 28096223